CLINICAL TRIAL: NCT01838447
Title: Prevention of Post-Cardiac Surgery Vitamin D Deficiency in Children With Congenital Heart Disease: A Pilot Dose Evaluation Randomized Controlled Trial
Brief Title: Prevention of Vitamin D Deficiency Following Pediatric CHD Surgery: a Phase II Dose Evaluation Randomized Controlled Trial Comparing Usual Care With a High Dose Pre-operative Supplementation Regimen Based on the Institute of Medicine Daily Upper Tolerable Intake Level
Acronym: HICCUPS 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Ottawa Hospital (Other); McGill University (Other); Children's University Hospital, Ireland (Other); Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, James Dayre McNally, Dr. James Dayre McNally, Pediatric Intensivist, Department of Pediatrics, CHEO, Associate Investigator, CHEO Research Institute, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VITAMINDINCHD-01
Record Dates: First submitted 2013-04-11; First posted 2013-04-24 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-05

CONDITIONS: Vitamin D Deficiency; Thoracic Surgery; Pediatric Disorders; Heart Defects, Congenital
Keywords: Vitamin D; Congenital Heart Disease; Cardiac Surgery; Pediatrics; Phase II Clinical Trial
MeSH Terms: conditions — Vitamin D Deficiency; Heart Defects, Congenital | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care group (No Intervention): This group will receive daily cholecalciferol (vitamin D3) based on the Adequate Intake (AI) for infants and the Recommended Dietary Allowance (RDA) for children over 1 year. Specific dose amounts are 400 IU per day for infants (0-1 year), and 600 IU per day for children between 1-17 years. Infants under 12 months of age who are formula fed will be given a placebo solution.
- High Dose Group (Experimental): This group will receive cholecalciferol (vitamin D3) based on the age-specific tolerable daily upper intake level (UL). Specific dose amounts are 1600 IU per day for infants (0-1 year), and 2400 IU per day for children between 1-17 years. Infants under 12 months of age who are formula fed will be given a dose of 1200 IU per day to account for vitamin D in formula.
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — The High Dose group is based on the age-specific UL. These doses were chosen to elevate 25OHD well above 50 nmol/L, while minimizing the risk of vitamin D toxicity (e.g. hypercalcemia, hypercalciuria)
  Other Names: Vitamin D3
  Arms: High Dose Group

SUMMARY:
Our research group has shown that almost all children with congenital heart disease (CHD) are vitamin D deficient following heart surgery. This work strongly suggests that the vitamin D intake presently recommended for healthy children, and also given to children with CHD, is inadequate to prevent vitamin D deficiency following surgery. Unfortunately, there have been no studies investigating any other vitamin D dose in children with heart disease. Recently, a higher dose of vitamin D intake has been approved (by the Institute of Medicine and Health Canada) and recent work on healthy children has shown it to be safe. The objective of this study is to determine whether this recently approved higher dose of vitamin D can safely reduce the number of children who are vitamin D deficient following surgery. This dose evaluation study will also evaluate whether it is possible to perform a large study (across Canada) to determine whether vitamin D supplementation can improve outcomes following surgery. It is hypothesized that a daily high dose vitamin D regimen, modeled on the Institute of Medicine daily upper tolerable intake level (UL), will significantly reduce vitamin D deficiency following CHD surgery, when compared with usual intake.

DETAILED DESCRIPTION:
1 - INTRODUCTION 1.1 Summary of problem CHD is a common condition with an estimated prevalence of 1 per 100 in the general population. A significant proportion of these pediatric patients require one or more corrective surgeries over their lifetime, leading to 15000 procedures per year in North America. Post-operatively, these patients suffer significant morbidities which may include a pronounced systemic inflammatory response, coagulopathy, respiratory failure, electrolyte disturbances, arrhythmia, myocardial dysfunction, kidney failure, infection and endocrine imbalances. Interventions that prevent or modulate post-operative pathophysiology may prevent illness, speed recovery and decrease chronic morbidity in this high risk pediatric population. Vitamin D is recognized as a pleiotropic hormone important for the functioning of multiple organ systems, including those central to critical illness pathophysiology. Recent research by our group and others has documented not only that 4 out of every 5 CHD patients have inadequate blood levels of vitamin D following surgery, but an association between immediate post-operative hormone levels and clinical course. Altogether, these findings and similar results in adult critical care and cardiac surgery populations, suggest that optimization of vitamin D status following CHD repair could lessen inflammation, reduce nosocomial infection and improve cardiac function. As an inexpensive medication (~$15/month) that is generally regarded as safe, vitamin D has the potential to be an ideal intervention for improving outcomes following CHD repair. Clinical trials will be required to determine whether elevation of pre-operative 25-hydroxyvitamin D (25OHD) and prevention of post-operative vitamin D deficiency improves the health of patients with CHD who require cardiac surgery.

1.2 - Gaps in current knowledge regarding vitamin D supplementation in CHD

The current body of knowledge suggests that optimization of vitamin D status prior to and following CHD repair could improve outcomes through reduced inflammation, fewer nosocomial infections and improved cardiac function. However, before these findings can be translated into clinical practice a number of unknowns must be addressed:

1. Evidence of benefit from interventional studies - As a unique and under-appreciated problem, there have been no interventional studies establishing that prevention of post-operative vitamin D deficiency improves clinical outcomes in CHD patients.
2. Lack of studies evaluating vitamin D dosing in the CHD population - Attempts to perform a large randomized control trial (RCT) would be premature as a dosing regimen that prevents post-operative vitamin D deficiency has not yet been identified. Moreover, there have been no vitamin D dosing studies or guidelines developed specific to the CHD population; presently children with CHD receive the same advice regarding supplementation as healthy children.
3. The safety of vitamin D doses above usual care has not been studied in the CHD population - Although it is tempting to extrapolate recent safety data from high dose vitamin D studies on healthy children to the CHD population, this may be inappropriate. CHD patients have unique metabolic demands, organ dysfunctions, and known and unknown genetic abnormalities that potentially make them more or less susceptible to vitamin D.

To begin addressing these knowledge gaps we will complete a pilot dose evaluation trial with the goal of identifying a supplementation regimen that safely prevents post-operative vitamin D deficiency.

2 - OBJECTIVES AND HYPOTHESIS 2.1 Hypothesis Pre-operative supplementation with a daily high dose vitamin D regimen, modeled on the Institute of Medicine (IOM) daily upper tolerable intake level (UL), will significantly reduce vitamin D deficiency following CHD surgery, when compared with usual intake.

2.2 Study objectives Primary study objective: In pediatric patients with CHD, determine whether a pre-operative regimen of daily high dose vitamin D results in a significant reduction in post-operative vitamin D deficiency, when compared with usual care

Secondary study objectives:

1. Determine whether a pre-operative regimen of daily high dose vitamin D, compared with usual care, results in vitamin D related adverse events (hypercalcemia, hypercalciuria).
2. Determine whether a pre-operative regimen of daily high dose vitamin D, compared with usual care, improves established markers of vitamin D axis functioning (active hormone levels, cardiac function).
3. Determine the barriers and feasibility of an RCT evaluating whether vitamin D supplementation improves clinical outcomes in children who require CHD surgery.

3 - METHODOLOGY 3.1 Study design and rationale - We will perform a pilot double blind randomized controlled dose evaluation trial comparing the efficacy and safety of two vitamin D dosing regimens in the prevention of post-operative vitamin D deficiency in children undergoing surgery for CHD.

3.2 Proposed supplement doses (Interventions) to be tested and rationale - Treatment groups - The doses for evaluation have been modelled on the two age specific intake levels recommended by the IOM. Infants under 6 months of age in the high dose group will receive 600 IU/day more than the IOM recommended UL, while those between 6 and 12 months will receive 100 IU/day more than UL.

Usual care group will receive Adequate Intake (AI) for infants and Recommended Dietary Allowance (RDA) for children over 1 year. These doses were chosen by IOM to achieve blood 25OHD levels above 50 nmol/L in the majority of the healthy population.

High dose group is based on the age-specific UL. These doses were chosen to elevate 25OHD well above 50 nmol/L, while minimizing risk of vitamin D toxicity (e.g. hypercalcemia, hypercalciuria).

3.3 Anticipated pre- and post-operative 25OHD levels in the study arms - Given the 40% intra-operative decline, pre-operative levels above 90 nmol/L will be required to maintain post-operative levels above 50 nmol/L (the value at which sufficient substrate to synthesize the active metabolite is available). The ability of certain vitamin D intake levels to achieve this pre-operative value can be inferred from recently completed dosing studies on healthy children level. These studies, including one by co-investigator (Dr. Hope Weiler, McGill) have shown that usual care dosing for 2 to 3 months will achieve pre-operative levels of 90 nmol/L in only 40-50%. In contrast, studies evaluating doses approximating our higher daily intake level (1600 IU/day ) achieved mean 25OHD levels of 130 to 150 nmol/L; suggesting that 80% of CHD patients could achieve pre-operative levels of 90 nmol/L or above.

3.4 Study design details 3.4.2 Stratification: We anticipate that two months of daily consumption may be required to achieve target 25OHD levels. Participants will be stratified into whether or not they are expected to receive at least 8 weeks of study drug prior to surgery. This stratification should guarantee that an equal number of CHD patients who will not receive 8 weeks of oral dosing end up in both the high and low dose arms. We will further stratify by the age (under or over 1 year of age) 3.4.3 Randomization and allocation concealment: Computer software generated randomization will be performed. Given the expected recruitment (4 to 5 per month) and potential impact of season on 25OHD randomization will be performed in blocks (4 within each strata). Only the pharmacy staff will be aware which patients receive high and low dose.

3.4.4 Blinding: We will blind patients, families, investigators, hospital staff, and research personnel to treatment arm. The two interventions will be indistinguishable (vial, volume, color, taste, consistency and smell). Only the pharmacist will know the identity of the study drug administered to a specific patient. Blinding can be broken at the request of the clinical service.

3.4.5 Co-interventions: The study protocol will not protocolize co-interventions as the study is single centre and CHEO has protocols or standardized approaches to the common post-operative complications and adverse events.

3.5 Study procedures 3.5.1 Recruitment: Potentially eligible study participants will be identified in the ambulatory clinics (cardiology, cardiovascular) or inpatient wards (including pediatric intensive care and neonatal intensive care unit). CHD patients identified as requiring surgery and have or will be referred to the cardiovascular team for consultation may be provided a patient brochure directly by hospital staff or as part of the standard information package (mailed to outpatients). Caregivers (and children where appropriate) will be asked for permission to be approached about study participation by the research nurse/assistant.

3.5.2 Study drug distribution: Europharm has agreed to provide the study drug in the required concentrations, prepared in indistinguishable vials for blinding purposes. Pharmacy will administer study drug (based on randomization, participant age and whether the patient is breast or formula fed). Infants with CHD assigned to the usual care arm will be given a placebo (0 IU/mL) as they will receive usual (recommended) vitamin D intake as part of formula.

3.5.3 Frequency and duration of follow-up appointments Planned additional study appointments- There will be no additional appointments planned for study purposes. Patients may require additional appointments if research tests identify clinically relevant findings.

Planned additional study phone calls - Research study staff will call caregivers and participants (where applicable) every two to four weeks to encourage compliance and provide education.

3.5.4 Frequency of biological sample collection and metabolites measured Before initiation of study drug - Urine - After consent is obtained and the study participant is waiting for the pharmacy to prepare the study drug we will gather a urine sample for determination of calcium:creatinine ratios. Where developmentally appropriate the participants will be asked to provide urine into a container. Urine bags will be placed on younger children.

Blood - Neonates and other study participants (mainly inpatients) requiring surgery within 2 months of diagnosis and enrollment will have blood collected prior to (or within 2 days) of starting study supplement for determination of 25OHD. These patients will not have blood collected for research purposes again until they are taken to the operating room.

During period of study drug administration - Blood - For those study participants who will receive study drug for more than 6 months we will measure 25OHD and calcium at the time of clinically indicated blood-work during regularly scheduled cardiology or cardiovascular surgery (CVS) clinic appointments At time of standard pre-surgical blood work - All outpatient participants will have blood collected at the time of standard pre-surgical blood work in preparation for the operation (two to three weeks prior to surgery). The blood will be sent to the CHEO laboratory for measurement of 25OHD and ionized calcium. Once completed, results will be forwarded to safety officer and study investigator (sealed).

Intraoperative biological samples and measurements- Blood - All study participants will have 2 mL of blood collected in the operating room following anesthesia and intubation, but prior to skin incision and initiation of cardiopulmonary bypass. Blood will also be sent to the CHEO laboratory for pre-operative ionized calcium determination. Remaining sample will be aliquoted and stored at -80 degrees Celsius (oC).

Urine - All study participants will have urine collected after insertion of the urinary catheter. The sample will be sent to the CHEO laboratory for determination of calcium:creatinine ratio. Study results will not appear on the patient hospital chart, but will be labeled with the study identification (ID) number and forwarded to the study investigator and safety officer for review.

Post-operative biological samples and other study measurements Blood - All study participants will have 2 mL of blood collected following separation from cardiopulmonary bypass (at admission to PICU). Further study participants will have 2 mL of blood collected on post-operative days 1, 3, 5 and 10 in the PICU. Samples will be collected from arterial or central venous catheters at the time of clinically indicated blood work. If these catheters have been removed, blood will be collected at the time of clinically indicated venipuncture. If patients are discharged to the ward before the day 10 research sample is collected a discharge sample will be collected at the time of discharge and no further research blood will be gathered.

Urine - All study participants will have urine collected from the urinary catheter on the first post-operative day. The samples will be sent to the CHEO laboratory for determination of calcium and creatine concentrations.

Echocardiography - A comprehensive exam will be performed immediately post-operatively (standard of care) and on the first post-operative day by a trained technician or pediatric cardiologist.

Case report form

1. Questionnaire - On the day of surgery the research coordinator will collect the participant dairies and unused study supplement. Information will also be collected on prescribed medications, nutrition, and additional supplement use.
2. Operative details - The research assistant will extract detailed operative information, including: cardiac lesion type, surgery performed, Risk Adjusted Congenital Heart Surgery (RACHS) score, total fluid intake and output, blood product and fluid administration and loss, hypothermia, need for deep hypothermic circulatory arrest (duration), aortic cross clamp times, cardiopulmonary bypass (CPB) circuit volumes, CPB circuit constituents, CPB time, occurrence of intraoperative hyper or hypocalcemia, administration of parenteral calcium, need for catecholamines following separation from CPB, occurrence of intra-operative arrhythmias.
3. PICU course - Clinically relevant information on clinical course and organ dysfunction will be collected, including: death, extracorporeal membrane oxygenation (ECMO), PRISM illness severity, cardiovascular dysfunction (fluid bolus requirements, inotrope/catecholamine use, arrhythmia), renal dysfunction (urine output, creatinine measurements, need for dialysis), hypocalcemia and calcium administration, duration of mechanical ventilation and duration of PICU stay.

3.5.5 Other metabolites and measurements on research specimens Remaining research blood will be used for research purposes only (measurement of antimicrobial peptides, cytokines, nutritional markers).

4 -STUDY SAFETY MEASURES 4.1 Background on vitamin D safety and toxicity Acute vitamin D toxicity is characterized by hypercalcemia or hypercalciuria, with the classic symptoms directly attributable to these abnormalities. Acute toxicity is a rare event that occurs in the context of overdose (accidental or prescribed megadoses in the range of 300,000-600,000 IU). The risk of acute vitamin D toxicity with this study is remote as it would require consumption of more than one vial of study drug to meet doses (~150,000 IU) and blood 25OHD levels known to cause toxicity.

Vitamin D toxicity due to genetic susceptibility - Concern about the safety of daily high dose vitamin D supplementation dates back to the 1950's when a rise in idiopathic infantile hypercalcemia (IIH) coincided with the implementation of higher daily vitamin D intake (~4000 IU/day). This small epidemic lead to a decrease in recommended daily vitamin D intake to levels that could prevent rickets and hypocalcemic seizures (400 IU/day). It is now thought that most cases of IIH are due to rare genetic conditions (1:10000) that increase susceptibility to vitamin D. Of these, patients with William's syndrome can have CHD as part of the constellation of symptoms and the proposed project will exclude these individuals.

Lack of subacute/chronic toxicity with IOM high dose in healthy children - Given recent suggestions that higher vitamin D levels might protect against non-bone disease, the safety of vitamin D doses above usual care (400-600 IU/day) has been reconsidered. To address this question the American and Canadian governments had the IOM assemble a committee of experts to provide recommendations based upon a comprehensive review of literature. In the final IOM report an age specific daily upper tolerable intake level was provided that was intended to safely elevate 25OHD levels while avoiding toxicity. Recently two blinded RCTs have shown that vitamin D supplementation at and slightly above the IOM daily upper tolerable intake level does not cause hypercalcemia or hypercalcuria. It is important to acknowledge that the IOM recommendations are for healthy children and may not be applicable to children with CHD 4.2 Safety measures and clinically relevant research findings Pre-surgical 25OHD and ionized calcium levels -

To avoid vitamin D overdose, hypercalcemia and side effects we have selected a supplement level recently proven to be safe in healthy children and will target the period of high dose supplementation to 6 months, and no more than 12 months. Further, to avoid excessive vitamin D levels at time of surgery we will measure 25OHD and ionized calcium with the pre-surgical blood work (~3 weeks prior to surgery for outpatients who will receive many months of supplementation). These values will be determined through the CHEO laboratory with results forwarded to the study investigator and safety officer. Study participants with elevated blood calcium and/or vitamin D levels will be identified and contacted by the safety officer. Ionized calcium thresholds have been established. For 25OHD, although 500 nmol/L is generally considered the definitive toxicity threshold, we have chosen to intervene with 25OHD levels above 200 nmol/L as this value is supraphysiological and exceeds our study goal. The following details the actions that will be taken with abnormal values:

1. For 25OHD above 200 nmol/L with evidence of hypercalcemia (vitamin D toxicity): discontinue study drug immediately, repeat the values (fasting), and refer to endocrinology.
2. For 25OHD above 200 nmol/L without hypercalcemia: study drug will be reduced by 50% (c) For 25OHD above 250 nmol/L, without hypercalcemia: study drug will be discontinued (d) For hypercalcemia with 25OHD under 200 nmol/L: repeat the bloodwork (fasting) and refer to endocrinology Pre-surgical 25OHD and ionized calcium levels during period of study drug administration. For patients who will receive more than 6 months of study drug prior to surgery we will determine blood 25OHD and ionized calcium at the time of routine bloodwork at CVS and cardiology appointments (or hospitalizations) Post-operative blood calcium levels. Will be determined at multiple times following cardiac surgery and represents standard of care. Both hypo and hypercalcemia will be managed by the clinical team as required. Study participants with persistently elevated blood calcium levels (for more than two days, not explained by intravenous calcium administration) will be referred to endocrinology.

   Post-treatment, pre-operative elevated urine calcium:creatinine ratios - As prolonged exposure to hypercalciuria (> 3 months) could theoretically cause nephrocalcinosis we will have ultrasounds performed prior to hospital discharge on all patients with elevated immediate pre-operative urine calcium to creatinine ratios. Any study participant with nephrocalcinosis will be referred to the CHEO nephrology service for further assessment. It is important to note that with the exception of a decrease in vitamin D dose to minimal daily intake (will occur by default in all patients) there would be no additional treatment for nephrocalcinosis at this time. Dr. Geier has offered to see these patients at no expense.

   Post-operative elevated urine calcium:creatinine ratios - Urine calcium to creatinine ratios are not measured as part of standard medical care. Further no research is available to indicate the impact of CHD and operative procedures on acute post-surgical calcium excretion or long-term nephrocalcinosis risk. However, as this patient population is followed closely and nephrocalcinosis is rarely reported following CHD surgery (only one case series of 3 in the literature) it does not appear that these patients are at significant risk for nephrocalcinosis. However, the addition of higher doses of vitamin D could predispose to nephrocalcinosis given concurrent acute illness, immobilization and diuretic use. Therefore any patient with an elevated calcium: creatinine ratio (collected on the first post-operative day) will be referred to nephrology service. Again, Dr. Geier has offered to consult on these patients; he will repeat the calcium: creatinine ratio and decide upon further investigation.

   Participants that have study drug discontinued or decreased will be retained in the study, have peri-operative biological samples collected as outlined, and will be included in the analysis using intention to treat methodology.

   4.3 Study results of unclear clinical relevance 4.3.1 Post-operative vitamin D Low risk of elevated post-operative vitamin D - As described, vitamin D levels will be checked 2 to 3 weeks prior to surgery. For patients with even moderate elevations in 25OHD (above 200 nmol/L) study drug intake will be modified to ensure vitamin D levels do not exceed 250 nmol/L in any individual at the time of surgery. Given these pre-operative safety measures and the known 40% intraoperative drop, we anticipate that no study participant will have a vitamin D level above 250 nmol/L post-operatively. Even if a participant was to have unexpectedly high 25OHD value, no treatment would be initiated without evidence of hypercalcemia (note - patients with persistent post-operative hypercalcemia would be referred to endocrinology as outlined in section 4.1). Further, the management plan for a post-operative patient with 25OHD in excess of 200 nmol/L would be to discontinue high dose study supplement. As all study participants will discontinue study drug at time of surgery, any patient with elevated 25OHD will already be receiving the appropriate management.

   Unclear relevance of low post-operative Vitamin D - Observational studies suggest that low post-operative vitamin D contributes to a more protracted clinical course. However, it is presently unclear whether or how to acutely increase 25OHD in post-operative CHD patients as there is no intravenous form and the safety of single enteral megadoses of vitamin D (>100,000 IU) has not been proven in any diseased pediatric population. With the exception of those participants with endocrinology consults initiated (for hypercalcemia) all patients will be encouraged to continue with standard vitamin D supplementation following surgery (infants 400 IU, children 600 IU). This intake will gradually restore 25OHD above 50 nmol/L over a 2 to 3 month period.

   Given the above rationale there would be no benefit in determining 25OHD values at the time of active patient care. For this reason, immediate pre and post-operative blood will be collected and stored at -80 oC for batch determination of vitamin D metabolites.

   4.3.2 Elevated urine calcium:creatinine Background - There is a theoretical increased risk of hypercalciuria leading to nephrocalcinosis with high dose vitamin D supplementation. Although frequently discussed in the literature the association between vitamin D supplementation and nephrocalcinosis appears limited to two rare circumstances: a rare genetic disorder called vitamin D resistant rickets and cumulative vitamin D intake above 600,000 (over a few days or month).

   Pre-treatment urine calcium/creatinine ratios - Given the absence of good evidence supporting a link between low to moderate dose daily enteral vitamin D intake and hypercalciuria and nephrocalcinosis we have decided not to exclude patients from the study based on their pre-treatment urine calcium to creatinine ratio. The pretreatment values will be reported in the two treatment groups and will be used to determine whether CHD patients with high initial values are more likely to have elevated calcium:creatinine ratios at the time of surgery and/or evidence of nephrocalcinosis. This finding would result in exclusion of these patients from the subsequent multicenter phase III study.

   4.4 Data Safety Monitoring Board (DSMB) A DSMB will be set up for this trial. Study results will be analyzed after half of the participants (n=32) have completed all study procedures, including assay for 25OHD, ionized calcium and urine calcium:creatinine ratios. With the biochemistry and information on clinical adverse events the DSMB will determine whether it is safe to continue the pilot study.

   5 - ETHICAL REVIEW AND CONSIDERATIONS The proposed trial has been reviewed by the Research Ethics Board at the Children's Hospital of Eastern Ontario. Informed consent will be obtained from all parents and from patients (assent, where applicable). All participation will be entirely voluntary and parents/children will be informed that they are free to refuse to participate or withdraw consent at any time during the course of the study without jeopardizing the excellence of the care they receive by the cardiovascular surgery program at CHEO. All information will be kept confidential, will be accessible only by the study personnel and treating team, and will not be released to a third party.

   6 - SAMPLE SIZE DETERMINATION Primary objective - Based on our observational studies and findings from recent dose evaluation studies on healthy children we estimate that 40% of the usual care arm will have post-operative 25OHD levels above 50 nmol/L. Based on the 25OHD levels achieved with 1600 IU/day in recent studies on approximate IOM high dose in healthy children we anticipate that 80% of the high dose arm will have post-operative levels above 50 nmol/L. Therefore group sample sizes of 28 in both treatment arms will be required to achieve 80% power to detect a difference between the group proportions of 0.40. The test statistic used is the two-sided Fisher's exact test and the significance level of the test was targeted at 0.05. Assuming a 10% drop out rate, 62 patients (total) will be recruited.

   Comments on power for evaluating vitamin D related adverse outcomes - (1) Hypercalcemia - Our observational study (n=58) identified no cases of pre-operative or immediate post-operative hypercalcemia. With a baseline rate in the usual care arm between 0 and 10% our sample size would be sufficient to show a statistically significant difference between groups if the rate in the high dose arm exceeded 30%. (2) Hypercalciuria - Information on baseline rates of hypercalciuria prior to or following cardiac surgery with usual care vitamin D intake is not available. The proposed sample size would be sufficient to demonstrate a 35% difference in proportions if the baseline pre or post-operative rates were between 0 and 20%.

   7 - STATISTICAL ANALYSIS The analyses for both studies will be performed using Statistical Analysis System (SAS) software (Copyright SAS Institute Inc., Cary, North Carolina, USA) and a p-value less than 0.05 will be considered statistically significant.

   Descriptive statistics - Treatment groups will be described and compared using: (i) means with standard deviations or medians with inter-quartile range values for continuous variables or (ii) frequencies with percentages for categorical variables. Statistically significant differences will be determined using Chi-square and Fisher's exact tests for categorical variables, and t-tests or nonparametric tests (e.g. Wilcoxon) for continuous variables, as appropriate.

   Primary outcome - The primary analytical approach will be to evaluate all randomized patients in an intention to treat analysis. Differences in the primary outcome measure, proportion with 25OHD < 50 nmol/L, between the treatment groups will be evaluated using the Fisher's exact test. Logistic regression analysis will be used if important variables are unevenly distributed between groups. *We anticipate minimal missing data as over 95% of participants from the recently completed observational study had an immediate post-operative sample.

   Secondary outcomes - Secondary analyses will be evaluated between groups based on data type. Outcome measures that are continuous will be evaluated using the t-test, Wilcoxon sign rank test (where appropriate) or through linear regression analysis if important variables are not evenly distributed between groups. Binary secondary outcome measures (e.g. hypercalcemia, hypercalciuria) will be compared between the two treatment groups using Fisher's exact or Chi-square. For the analysis of outcomes measures that represent time to event (e.g. restoration of active hormone (1,25OH2D) levels to normal range, time to extubation, PICU length of stay) we will apply the log rank test. If randomization does not lead to equal distribution of important variables (e.g. weight) the analysis will be expanded to multiple regression modeling.

   Subgroup analysis - The well known pharmacology of enteral vitamin D dosing shows that at least 2 months of regular daily intake is required to build body stores and achieve steady state blood levels of vitamin D. Consequentially neonates or other infants enrolled into the study who require surgery within two months of birth or CHD diagnosis will be analyzed separately. Primary objective - Similar to the outpatient study the primary objective in this subgroup is to report the proportions (in the usual care and high dose groups) that are vitamin D deficient post-operatively. However, given that these participants will receive study drug for a very short period we anticipate that the proportion with 25OHD levels above 50 nmol/L will remain low in the high dose group. Our program goal at this stage is to identify a dosing regimen that prevent post-operative vitamin D deficiency in 75% of CHD patients. Given this goal, and an estimated prevalence of 15 to 35% we would need 12 neonates per group to generate a confidence interval that excludes 75%. As neonates represent 20% of all CHD surgeries, we anticipate that enrolling 62 total subjects will be sufficient.

   Feasibility - Most neonates with CHD who require cardiac surgery within the first few weeks of life have serious cardiac lesions that can limit enteral nutrition and medication delivery. Anticipating that most of these patients will not significantly elevate 25OHD levels with daily enteral intake at IOM high dose this study will provide important information on the willingness of health care providers to provide enteral study drug. This information will allow us to consider alternative dosing regimen for future studies based on single or divided representing one or more months worth of daily dosing (e.g. 5-10,000 IU/kg).

   8 - STUDY TEAM AND MANAGEMENT The principal investigator (DM) and co-investigator (KM) will be responsible for supervision of the study. The research nurse and assistant(s) will be responsible for participant recruitment and day-to-day management. The Clinical Research Unit at the CHEO Research Institute which will provide administrative and data management support. Co-investigator, Dean Fergusson will assist with methodology, analysis, and interpretation

ELIGIBILITY:
Inclusion Criteria:

* Newborn (corrected gestational age between 36 weeks) up to 18 years
* Has CHD that will require surgery within the next 12 months
* CHD requiring surgical intervention with cardiopulmonary bypass

Exclusion Criteria:

* Born at less than 32 weeks gestational age
* Corrected gestational age of less than 36 weeks
* Cardiac or gastrointestinal disease preventing enteral feeds or drug administration prior to surgery
* Patient has confirmed or suspected Williams syndrome
* Proposed surgery to take place at another centre (outside of CHEO)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D McNally, M.D., Ph.D., Principal Investigator — Children's Hospital of Eastern Ontario; Kusum Menon, M.D., Study Chair — Children's Hospital of Eastern Ontario; Lauralyn McIntyre, M.D., Study Chair — Ottawa Hospital; Dermot R Doherty, M.B., B.Ch., Study Chair — Temple Street Children's University Hospital Dublin and University College; Dean Ferguson, Ph.D., Study Chair — Ottawa Hospital Research Institute; Hope Weiler, Ph.D., Study Chair — McGill University
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Background] McNally JD, Menon K, Chakraborty P, Fisher L, Williams KA, Al-Dirbashi OY, Doherty DR; Canadian Critical Care Trials Group. The association of vitamin D status with pediatric critical illness. Pediatrics. 2012 Sep;130(3):429-36. doi: 10.1542/peds.2011-3059. Epub 2012 Aug 6. PMID 22869837
- [Background] Thacher TD, Clarke BL. Vitamin D insufficiency. Mayo Clin Proc. 2011 Jan;86(1):50-60. doi: 10.4065/mcp.2010.0567. PMID 21193656
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Wandrup J. Critical analytical and clinical aspects of ionized calcium in neonates. Clin Chem. 1989 Oct;35(10):2027-33. PMID 2676238
- [Background] Loughead JL, Mimouni F, Tsang RC. Serum ionized calcium concentrations in normal neonates. Am J Dis Child. 1988 May;142(5):516-8. doi: 10.1001/archpedi.1988.02150050054030. PMID 3358391
- [Background] Roberts KE. Pediatric fluid and electrolyte balance: critical care case studies. Crit Care Nurs Clin North Am. 2005 Dec;17(4):361-73, x. doi: 10.1016/j.ccell.2005.07.006. PMID 16344206
- [Background] Sargent JD, Stukel TA, Kresel J, Klein RZ. Normal values for random urinary calcium to creatinine ratios in infancy. J Pediatr. 1993 Sep;123(3):393-7. doi: 10.1016/s0022-3476(05)81738-x. PMID 8355114
- [Background] Safarinejad MR. Urinary mineral excretion in healthy Iranian children. Pediatr Nephrol. 2003 Feb;18(2):140-4. doi: 10.1007/s00467-002-1020-1. Epub 2002 Dec 21. PMID 12579403
- [Background] Erol I, Buyan N, Ozkaya O, Sahin F, Beyazova U, Soylemezoglu O, Hasanoglu E. Reference values for urinary calcium, sodium and potassium in healthy newborns, infants and children. Turk J Pediatr. 2009 Jan-Feb;51(1):6-13. PMID 19378884
- [Background] Matos V, van Melle G, Boulat O, Markert M, Bachmann C, Guignard JP. Urinary phosphate/creatinine, calcium/creatinine, and magnesium/creatinine ratios in a healthy pediatric population. J Pediatr. 1997 Aug;131(2):252-7. doi: 10.1016/s0022-3476(97)70162-8. PMID 9290612
- [Background] Matos V, Van Melle G, Werner D, Bardy D, Guignard JP. Urinary oxalate and urate to creatinine ratios in a healthy pediatric population. Am J Kidney Dis. 1999 Aug;34(2):e1. doi: 10.1053/AJKD034000e6. PMID 10430995
- [Background] Hata TR, Kotol P, Jackson M, Nguyen M, Paik A, Udall D, Kanada K, Yamasaki K, Alexandrescu D, Gallo RL. Administration of oral vitamin D induces cathelicidin production in atopic individuals. J Allergy Clin Immunol. 2008 Oct;122(4):829-831. doi: 10.1016/j.jaci.2008.08.020. No abstract available. PMID 19014773
- [Background] Gombart AF, Borregaard N, Koeffler HP. Human cathelicidin antimicrobial peptide (CAMP) gene is a direct target of the vitamin D receptor and is strongly up-regulated in myeloid cells by 1,25-dihydroxyvitamin D3. FASEB J. 2005 Jul;19(9):1067-77. doi: 10.1096/fj.04-3284com. PMID 15985530
- [Background] Liu PT, Stenger S, Tang DH, Modlin RL. Cutting edge: vitamin D-mediated human antimicrobial activity against Mycobacterium tuberculosis is dependent on the induction of cathelicidin. J Immunol. 2007 Aug 15;179(4):2060-3. doi: 10.4049/jimmunol.179.4.2060. PMID 17675463
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827
- [Background] Holmlund-Suila E, Viljakainen H, Hytinantti T, Lamberg-Allardt C, Andersson S, Makitie O. High-dose vitamin d intervention in infants--effects on vitamin d status, calcium homeostasis, and bone strength. J Clin Endocrinol Metab. 2012 Nov;97(11):4139-47. doi: 10.1210/jc.2012-1575. Epub 2012 Aug 29. PMID 22933541
- [Background] Gallo S. et al. Supplementation with oral vitamin D3 (400 IU/day) supports plasma levels of 25-hydroxyvitamin D of 50nmol/L but higher intakes required to reach 75 nmol/L in breastfed infants. Canadian Paediatric Society Annual Conference, 2012.
- [Background] Gallo S, Trussler K, Vanstone C, Rodd C, Weiler H. New ionized calcium values for newborn infants. American Society for Bone Research, 2008.
- [Background] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Background] Brix-Christensen V. The systemic inflammatory response after cardiac surgery with cardiopulmonary bypass in children. Acta Anaesthesiol Scand. 2001 Jul;45(6):671-9. doi: 10.1034/j.1399-6576.2001.045006671.x. PMID 11421823
- [Background] Gazit AZ, Huddleston CB, Checchia PA, Fehr J, Pezzella AT. Care of the pediatric cardiac surgery patient--part 1. Curr Probl Surg. 2010 Mar;47(3):185-250. doi: 10.1067/j.cpsurg.2009.11.006. No abstract available. PMID 20159189
- [Background] McEwan A. Aspects of bleeding after cardiac surgery in children. Paediatr Anaesth. 2007 Dec;17(12):1126-33. doi: 10.1111/j.1460-9592.2007.02265.x. No abstract available. PMID 17986030
- [Background] Dyke PC 2nd, Yates AR, Cua CL, Hoffman TM, Hayes J, Feltes TF, Springer MA, Taeed R. Increased calcium supplementation is associated with morbidity and mortality in the infant postoperative cardiac patient. Pediatr Crit Care Med. 2007 May;8(3):254-7. doi: 10.1097/01.PCC.0000260784.30919.9E. PMID 17417127
- [Background] Lee P. Vitamin D metabolism and deficiency in critical illness. Best Pract Res Clin Endocrinol Metab. 2011 Oct;25(5):769-81. doi: 10.1016/j.beem.2011.03.001. PMID 21925077
- [Background] Lee P, Eisman JA, Center JR. Vitamin D deficiency in critically ill patients. N Engl J Med. 2009 Apr 30;360(18):1912-4. doi: 10.1056/NEJMc0809996. No abstract available. PMID 19403914
- [Background] Amrein K, Venkatesh B. Vitamin D and the critically ill patient. Curr Opin Clin Nutr Metab Care. 2012 Mar;15(2):188-93. doi: 10.1097/MCO.0b013e32834f0027. PMID 22186356
- [Background] Graham EM, Taylor SN, Zyblewski SC, Wolf B, Bradley SM, Hollis BW, McGowan FX Jr, Atz AM. Vitamin D status in neonates undergoing cardiac operations: relationship to cardiopulmonary bypass and association with outcomes. J Pediatr. 2013 Apr;162(4):823-6. doi: 10.1016/j.jpeds.2012.10.013. Epub 2012 Nov 10. PMID 23149171
- [Background] Lucidarme O, Messai E, Mazzoni T, Arcade M, du Cheyron D. Incidence and risk factors of vitamin D deficiency in critically ill patients: results from a prospective observational study. Intensive Care Med. 2010 Sep;36(9):1609-11. doi: 10.1007/s00134-010-1875-8. Epub 2010 Apr 7. No abstract available. PMID 20373095
- [Background] McKinney JD, Bailey BA, Garrett LH, Peiris P, Manning T, Peiris AN. Relationship between vitamin D status and ICU outcomes in veterans. J Am Med Dir Assoc. 2011 Mar;12(3):208-11. doi: 10.1016/j.jamda.2010.04.004. PMID 21333923
- [Background] Higgins DM, Wischmeyer PE, Queensland KM, Sillau SH, Sufit AJ, Heyland DK. Relationship of vitamin D deficiency to clinical outcomes in critically ill patients. JPEN J Parenter Enteral Nutr. 2012 Nov;36(6):713-20. doi: 10.1177/0148607112444449. Epub 2012 Apr 20. PMID 22523178
- [Background] Braun A, Chang D, Mahadevappa K, Gibbons FK, Liu Y, Giovannucci E, Christopher KB. Association of low serum 25-hydroxyvitamin D levels and mortality in the critically ill. Crit Care Med. 2011 Apr;39(4):671-7. doi: 10.1097/CCM.0b013e318206ccdf. PMID 21242800
- [Background] Braun AB, Gibbons FK, Litonjua AA, Giovannucci E, Christopher KB. Low serum 25-hydroxyvitamin D at critical care initiation is associated with increased mortality. Crit Care Med. 2012 Jan;40(1):63-72. doi: 10.1097/CCM.0b013e31822d74f3. PMID 21926604
- [Background] Zittermann A, Schleithoff SS, Gotting C, Fuchs U, Kuhn J, Kleesiek K, Tenderich G, Koerfer R. Calcitriol deficiency and 1-year mortality in cardiac transplant recipients. Transplantation. 2009 Jan 15;87(1):118-24. doi: 10.1097/TP.0b013e31818c2708. PMID 19136901
- [Background] Matthews LR, Ahmed Y, Wilson KL, Griggs DD, Danner OK. Worsening severity of vitamin D deficiency is associated with increased length of stay, surgical intensive care unit cost, and mortality rate in surgical intensive care unit patients. Am J Surg. 2012 Jul;204(1):37-43. doi: 10.1016/j.amjsurg.2011.07.021. Epub 2012 Feb 10. PMID 22325335
- [Background] Madden K, Feldman HA, Smith EM, Gordon CM, Keisling SM, Sullivan RM, Hollis BW, Agan AA, Randolph AG. Vitamin D deficiency in critically ill children. Pediatrics. 2012 Sep;130(3):421-8. doi: 10.1542/peds.2011-3328. Epub 2012 Aug 6. PMID 22869836
- [Background] Borgermann J, Lazouski K, Kuhn J, Dreier J, Schmidt M, Gilis-Januszewski T, Knabbe C, Gummert JF, Zittermann A. 1,25-Dihydroxyvitamin D fluctuations in cardiac surgery are related to age and clinical outcome*. Crit Care Med. 2012 Jul;40(7):2073-81. doi: 10.1097/CCM.0b013e31824e8c42. PMID 22584760
- [Background] Pierpont ME, Basson CT, Benson DW Jr, Gelb BD, Giglia TM, Goldmuntz E, McGee G, Sable CA, Srivastava D, Webb CL; American Heart Association Congenital Cardiac Defects Committee, Council on Cardiovascular Disease in the Young. Genetic basis for congenital heart defects: current knowledge: a scientific statement from the American Heart Association Congenital Cardiac Defects Committee, Council on Cardiovascular Disease in the Young: endorsed by the American Academy of Pediatrics. Circulation. 2007 Jun 12;115(23):3015-38. doi: 10.1161/CIRCULATIONAHA.106.183056. Epub 2007 May 22. PMID 17519398
- [Background] Kobrynski LJ, Sullivan KE. Velocardiofacial syndrome, DiGeorge syndrome: the chromosome 22q11.2 deletion syndromes. Lancet. 2007 Oct 20;370(9596):1443-52. doi: 10.1016/S0140-6736(07)61601-8. PMID 17950858
- [Background] Markestad T, Hesse V, Siebenhuner M, Jahreis G, Aksnes L, Plenert W, Aarskog D. Intermittent high-dose vitamin D prophylaxis during infancy: effect on vitamin D metabolites, calcium, and phosphorus. Am J Clin Nutr. 1987 Oct;46(4):652-8. doi: 10.1093/ajcn/46.4.652. PMID 3499065
- [Background] Schlingmann KP, Kaufmann M, Weber S, Irwin A, Goos C, John U, Misselwitz J, Klaus G, Kuwertz-Broking E, Fehrenbach H, Wingen AM, Guran T, Hoenderop JG, Bindels RJ, Prosser DE, Jones G, Konrad M. Mutations in CYP24A1 and idiopathic infantile hypercalcemia. N Engl J Med. 2011 Aug 4;365(5):410-21. doi: 10.1056/NEJMoa1103864. Epub 2011 Jun 15. PMID 21675912
- [Background] Jenkins KJ, Gauvreau K, Newburger JW, Spray TL, Moller JH, Iezzoni LI. Consensus-based method for risk adjustment for surgery for congenital heart disease. J Thorac Cardiovasc Surg. 2002 Jan;123(1):110-8. doi: 10.1067/mtc.2002.119064. PMID 11782764
- [Background] Gordon CM, Williams AL, Feldman HA, May J, Sinclair L, Vasquez A, Cox JE. Treatment of hypovitaminosis D in infants and toddlers. J Clin Endocrinol Metab. 2008 Jul;93(7):2716-21. doi: 10.1210/jc.2007-2790. Epub 2008 Apr 15. PMID 18413426
- [Background] Pollack MM, Patel KM, Ruttimann UE. The Pediatric Risk of Mortality III--Acute Physiology Score (PRISM III-APS): a method of assessing physiologic instability for pediatric intensive care unit patients. J Pediatr. 1997 Oct;131(4):575-81. doi: 10.1016/s0022-3476(97)70065-9. PMID 9386662
- [Background] Cesur Y, Caksen H, Gundem A, Kirimi E, Odabas D. Comparison of low and high dose of vitamin D treatment in nutritional vitamin D deficiency rickets. J Pediatr Endocrinol Metab. 2003 Oct-Nov;16(8):1105-9. doi: 10.1515/jpem.2003.16.8.1105. PMID 14594170
- [Background] Soliman AT, El-Dabbagh M, Adel A, Al Ali M, Aziz Bedair EM, Elalaily RK. Clinical responses to a mega-dose of vitamin D3 in infants and toddlers with vitamin D deficiency rickets. J Trop Pediatr. 2010 Feb;56(1):19-26. doi: 10.1093/tropej/fmp040. Epub 2009 Jun 8. PMID 19506025
- [Background] Zeghoud F, Ben-Mekhbi H, Djeghri N, Garabedian M. Vitamin D prophylaxis during infancy: comparison of the long-term effects of three intermittent doses (15, 5, or 2.5 mg) on 25-hydroxyvitamin D concentrations. Am J Clin Nutr. 1994 Sep;60(3):393-6. doi: 10.1093/ajcn/60.3.393. PMID 8074071
- [Background] Tau C, Ciriani V, Scaiola E, Acuna M. Twice single doses of 100,000 IU of vitamin D in winter is adequate and safe for prevention of vitamin D deficiency in healthy children from Ushuaia, Tierra Del Fuego, Argentina. J Steroid Biochem Mol Biol. 2007 Mar;103(3-5):651-4. doi: 10.1016/j.jsbmb.2006.12.027. Epub 2007 Jan 25. PMID 17257830
- [Background] Oliveri B, Cassinelli H, Mautalen C, Ayala M. Vitamin D prophylaxis in children with a single dose of 150000 IU of vitamin D. Eur J Clin Nutr. 1996 Dec;50(12):807-10. PMID 8968701
- [Background] MITCHELL RG. Idiopathic hypercalcaemia of infants. Proc Nutr Soc. 1958;17(1):71-4. doi: 10.1079/pns19580013. No abstract available. PMID 13542614
- [Background] MITCHELL RG. The prognosis in idiopathic hypercalcaemia of infants. Arch Dis Child. 1960 Aug;35(182):383-8. doi: 10.1136/adc.35.182.383. No abstract available. PMID 13771357
- [Background] LIGHTWOOD R, STAPLETON T. Idiopathic hypercalcaemia in infants. Lancet. 1953 Aug 1;265(6779):255-6. doi: 10.1016/s0140-6736(53)90187-1. No abstract available. PMID 13070618
- [Background] BONGIOVANNI AM, EBERLEIN WR, JONES IT. Idiopathic hypercalcemia of infancy, with failure to thrive; report of three cases, with a consideration of the possible etiology. N Engl J Med. 1957 Nov 14;257(20):951-8. doi: 10.1056/NEJM195711142572001. No abstract available. PMID 13483867
- [Background] RHANEY K, MITCHELL RG. Idiopathic hypercalcaemia of infants. Lancet. 1956 Jun 30;270(6931):1028-32. doi: 10.1016/s0140-6736(56)90798-x. No abstract available. PMID 13333114
- [Background] Vieth R. Vitamin D toxicity, policy, and science. J Bone Miner Res. 2007 Dec;22 Suppl 2:V64-8. doi: 10.1359/jbmr.07s221. PMID 18290725
- [Background] Ammenti A, Pelizzoni A, Cecconi M, Molinari PP, Montini G. Nephrocalcinosis in children: a retrospective multi-centre study. Acta Paediatr. 2009 Oct;98(10):1628-31. doi: 10.1111/j.1651-2227.2009.01401.x. Epub 2009 Jul 1. PMID 19572991
- [Background] Ronnefarth G, Misselwitz J. Nephrocalcinosis in children: a retrospective survey. Members of the Arbeitsgemeinschaft fur padiatrische Nephrologie. Pediatr Nephrol. 2000 Sep;14(10-11):1016-21. doi: 10.1007/s004670050065. PMID 10975319
- [Background] Moncrieff MW, Chance GW. Nephrotoxic effect of vitamin D therapy in vitamin D refractory rickets. Arch Dis Child. 1969 Oct;44(237):571-9. doi: 10.1136/adc.44.237.571. No abstract available. PMID 5350034
- [Background] Mantan M, Bagga A, Virdi VS, Menon S, Hari P. Etiology of nephrocalcinosis in northern Indian children. Pediatr Nephrol. 2007 Jun;22(6):829-33. doi: 10.1007/s00467-006-0425-7. Epub 2007 Feb 7. PMID 17285294
- [Background] Atabek ME, Pirgon O, Sert A. Oral alendronate therapy for severe vitamin D intoxication of the infant with nephrocalcinosis. J Pediatr Endocrinol Metab. 2006 Feb;19(2):169-72. doi: 10.1515/jpem.2006.19.2.169. PMID 16562591
- [Background] Alon US. Nephrocalcinosis. Curr Opin Pediatr. 1997 Apr;9(2):160-5. PMID 9204244
- [Background] Hathcock JN, Shao A, Vieth R, Heaney R. Risk assessment for vitamin D. Am J Clin Nutr. 2007 Jan;85(1):6-18. doi: 10.1093/ajcn/85.1.6. PMID 17209171
- [Background] Committee on Genetics. American Academy of Pediatrics: Health care supervision for children with Williams syndrome. Pediatrics. 2001 May;107(5):1192-204. PMID 11331709
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] McNally JD, O'Hearn K, Fergusson DA, Lougheed J, Doherty DR, Maharajh G, Weiler H, Jones G, Khamessan A, Redpath S, Geier P, McIntyre L, Lawson ML, Girolamo T, Menon K; Canadian Critical Care Trials Group. Prevention of post-cardiac surgery vitamin D deficiency in children with congenital heart disease: a pilot feasibility dose evaluation randomized controlled trial. Pilot Feasibility Stud. 2020 Oct 22;6:159. doi: 10.1186/s40814-020-00700-3. eCollection 2020. PMID 33110622
- [Derived] McNally JD, O'Hearn K, Lawson ML, Maharajh G, Geier P, Weiler H, Redpath S, McIntyre L, Fergusson D, Menon K; Canadian Critical Care Trials Groups. Prevention of vitamin D deficiency in children following cardiac surgery: study protocol for a randomized controlled trial. Trials. 2015 Sep 9;16:402. doi: 10.1186/s13063-015-0922-8. PMID 26353829

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care Group | High Dose Group
Started | 22 | 24
Completed | 20 | 21
Not Completed | 2 | 3
Not completed — Change in surgical plan | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Group | High Dose Group | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 3.8 [0.8 to 35.6] | 4.6 [1.0 to 45.6] | 4.3 [1.1 to 37.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 13 | 10 | 23
Weight (kg) [Median (Inter-Quartile Range); unit: kilograms] | 5.8 [3.6 to 12.9] | 5.4 [4.2 to 13.4] | 5.7 [4.1 to 13.2]
RACHS Score [Median (Inter-Quartile Range); unit: units on a scale] — The Risk Adjustment in Congenital Heart Surgery (RACHS) allows a detailed understanding of differences in mortality among pediatric patients who are undergoing surgery for congenital heart disease (CHD). Patients are assigned to to one of 6 risk categories (Risk Category 1 to Risk Category 6) based on the type of cardiac procedures. The risk categories group cardiac procedures with similar risks for in-hospital death together. A higher risk category means a higher risk of in-hospital death.
  units on a scale | 3 [2 to 4] | 2 [2 to 3] | 3 [2 to 3]
Other active medical condition [Count of Participants; unit: Participants] | 7 | 7 | 14
Surgery season [Count of Participants; unit: Participants]
  Winter | 5 | 6 | 11
  Spring | 2 | 3 | 5
  Summer | 8 | 6 | 14
  Fall | 5 | 6 | 11
Ethnicity [Count of Participants; unit: Participants]
  Caucasian | 14 | 14 | 28
  Aboriginal | 1 | 1 | 2
  Oriental | 3 | 0 | 3
  African/West Indian | 1 | 2 | 3
  Unknown/Other | 1 | 4 | 5
Expected Duration to Surgery at Time of Enrolment [Count of Participants; unit: Participants]
  <2 months | 18 | 18 | 36
  >2 months | 2 | 3 | 5
Type of Feeding in Children <1 year [Count of Participants; unit: Participants] — Population: Type of feeding is described for the sub-set of study participants who were <1 year of age at the time of randomization
  Participants
    number analyzed (Participants) | 12 | 12 | 24
    Breast fed | 9 | 10 | 19
    Formula fed | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Blood 25 Hydroxyvitamin D (25OHD) Concentrations
Description: Blood 25OHD will be measured to determine vitamin D deficiency, with a concentration below 50 nmol/L used to define deficiency. A PICU admission blood sample could not be obtained for one patient in the Usual Care Group and one patient in the High Dose Group, thus the total number analyzed differs from the full sample size.
Time Frame: 1 day (On admission to the pediatric intensive care unit (PICU) following CHD surgery)
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Usual Care Group | High Dose Group
Number analyzed (Participants) | 19 | 20
nmol/L | 34.8 (12.0) | 52.0 (23.3)

2. Secondary Outcome: Number of Participants With Hypercalcemia as a Vitamin D Related Adverse Event
Description: Hypercalcemia will be defined as an ionized calcium level above 1.40 mmol/L; or above 1.45 mmol/L for children under 8 weeks. Hypercalcemia will be evaluated in blood collected immediately before CHD surgery and throughout the post-operative course (measurements are standard of care).
Time Frame: Immediately before surgery, on admission to the PICU following CHD surgery, and on post-operative days 1,3,5 & 10
Measure: Number; unit: No. participants with hypercalcemia
Arm/Group | Usual Care Group | High Dose Group
Number analyzed (Participants) | 20 | 21
No. participants with hypercalcemia | 0 | 0

3. Secondary Outcome: Number of Participants With Hypercalciuria
Description: Hypercalciuria will be identified using calcium:creatinine ratios defined using age-specific norms and thresholds.
Time Frame: Immediately before surgery, on admission to the PICU following CHD surgery, and on the first post-operative day
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | High Dose Group
Number analyzed (Participants) | 20 | 21
Participants
  Enrolment | 1 | 0
  Intra-operative | 3 | 4
  Post-Operative Day 1 | 2 | 1

4. Secondary Outcome: Vitamin D Parathyroid Renal Axis Function Through Changes in Blood 1,25-dihydroxycholecalciferol
Description: Impaired vitamin D axis function will be defined as an inability to restore and maintain active hormone levels in the normal range following surgery after the first post-operative day
Time Frame: Immediately before surgery, on admission to the PICU following CHD surgery, and on post-operative days 1,3,5 & 10
Population: Data cannot be reported. Data was not collected.
Arm/Group | Usual Care Group | High Dose Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Changes in Cathelicidin as Measure of Innate Immune Function
Time Frame: Immediately before surgery, on admission to the PICU following CHD surgery, and on post-operative days 1,3,5 & 10
Population: This data cannot be reported. Data was not collected.
Arm/Group | Usual Care Group | High Dose Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Post-operative PICU Catecholamine Requirements
Description: Primarily, post-operative catecholamine requirements during the PICU admission will be evaluated as a dichotomous variable (yes/no). If a difference is noted in the primary analysis, inotrope requirements will be determined using the inotrope score, evaluated as the maximum score and in a time to event approach (off all inotropes, score of zero)
Time Frame: At any point between PICU admission and discharge, an average length of 5-7 days and not longer than 60 days
Population: Only the primary analysis (post-operative catecholamine requirements during the PICU admission will be evaluated as a dichotomous variable (yes/no)) was completed. Since there was not a significant difference between groups for this variable, we did not perform the secondary analysis (inotrope score).
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | High Dose Group
Number analyzed (Participants) | 20 | 21
Participants | 15 | 11

7. Secondary Outcome: Cardiovascular Function Through an Echocardiogram
Description: The post-operative day 1 echocardiogram will be used to evaluate for differences in cardiovascular function between study arms.
Time Frame: Post-operative day 1
Population: This data cannot be reported. Data was not collected.
Arm/Group | Usual Care Group | High Dose Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of study enrollment until post-operative hospital discharge or 90 days following surgery for congenital heart disease (whichever occurred first)
Description: Transient hypercalciuria without clinical symptoms was monitored but was not considered an adverse event. A priori, only persistent hypercalciuria with clinical symptoms was classified as an adverse event.
Arm/Group | Usual Care Group | High Dose Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No